CLINICAL TRIAL: NCT05992025
Title: Randomized Controlled Trial: Digital Phenotyping and Lifestyle Intervention in Patients with Myasthenia Gravis to Reduce Fatigue
Brief Title: Digital Phenotyping and Lifestyle Intervention in Patients with Myasthenia Gravis
Acronym: DIG-MG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-01455-01
Record Dates: First submitted 2023-06-07; First posted 2023-08-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Myasthenia Gravis
Keywords: lifestyle intervention; fatigue; OURA; physical activity
MeSH Terms: conditions — Myasthenia Gravis; Fatigue; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled trial, parallel-group design
Who Masked: Outcomes Assessor
Masking Description: The statistician responsible for the outcome analysis will be blinded as to what intervention each group has had.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Observation (No Intervention): Observation with the OURA ring and no digital meetings. The participants are offered delayed randomization after the study period. This group's outcome from the delayed randomization will be for the exploratory analysis, i.e., not in the primary analysis.
- Physical activity (Experimental): 12 weeks of physical activity guidance with short discussions via online group meetings according to a schedule. The participants in this arm will conduct moderate-intensity exercises for at least 150 minutes per week. Brisk walks are the primary choice of activity; alternatively, swimming, cycling, or dancing to the physical exertion according to the Borg scale can be performed.
  Interventions: Behavioral: Physical activity
- Sleep hygiene intervention (Active Comparator): 12 weeks of sleep exercises. The lifestyle intervention of sleep will be delivered via an online group, with recommended home practices between sessions. Topics covered will include sleep education, sleep hygiene, and practices to improve sleep quality.
  Interventions: Behavioral: Sleep hygiene

INTERVENTIONS:
Behavioral: Physical activity — Intervention with physical activity more than 150 minutes of medium to high intensity per week.
  Arms: Physical activity
Behavioral: Sleep hygiene — Intervention with sleep hygiene to optimize sleep duration and quality.
  Arms: Sleep hygiene intervention

SUMMARY:
Myasthenia Gravis (MG) is a chronic autoimmune neurological disorder where an antibody attack of muscle receptors causes fatigable skeletal muscle weakness. In addition to fatigue, several MG patients experience general fatigue. Small supervised studies during 12 weeks of physical exercise interventions have indicated safety and beneficial neuromuscular outcomes in MG patients. Longer and unsupervised studies are required to obtain guidelines for physical activity in MG patients. Further, the development of smart rings enables remote digital supervision of physical activity, sleep, and biological parameters such as heart frequency, number of steps, and temperature. These parameters could add to the lack of biomarkers in MG. The project design is a randomized controlled trial with a lifestyle intervention to improve fatigue in the autoimmune neuromuscular disease Myasthenia Gravis (MG). The intervention includes digital group counseling regarding physical activity, sleep, general health, and digital follow-up with a "smart ring" (OURA).

DETAILED DESCRIPTION:
The cohort is Myasthenia Gravis (MG) patients in Sweden. The primary research question is: can digital lifestyle intervention in an online-group format improve fatigue as measured by MG-ADL in MG patients by at least 30%? Secondary research question: can lifestyle intervention improve fatigue as measured by FSS in MG by at least 30%?

The primary outcome measure is MG-ADL; the secondary outcome measures include general fatigue (fatigue severity scale and Chalder´s fatigue scale). Exploratory outcome measures include OURA-ring-based markers, including heart rate variability, temperature fluctuations, and sleep and activity parameters. These will be collected throughout the entire study period for 30 weeks.

Analysis of serum biomarkers miR-150-5p and miR-30e-5p and inflammatory proteins found upregulated in MG will be included. Clinical data at baseline: antibody status, electrophysiology, MG Composite Scale (MGC), and clinical data at follow-up visits (medications, MGC), etc., are extracted from the medical charts and the Swedish MG registry

Inclusion criteria:

* An MG diagnosis for at least six months before entry into the study.
* Both patients with ocular and generalized MG are allowed to participate.
* For practical reasons, participants need to understand Swedish.

Exclusion criteria:

* Participation in another clinical trial in the past 6 months.
* Disease duration less than 6 months.
* Contraindications to physical activity: unstable coronary syndrome or myocardial infarction within the preceding three months, respiratory failure (vital capacity < 70% predicted value) or cardiac failure (ejection fraction < 50% predicted value), concomitant neuromuscular diseases, disabling rheumatological disease (> 80% disability on the Barthel scale), chronic pain or disabling orthopedic conditions, hospitalization in the last three months for a serious medical or surgical condition, anemia (hematocrit < 30%), stroke within the previous year.
* MG patients already performing a moderate-intensity physical activity of 150min or more per week, i.e., one of the target interventions.
* Pregnancy.

Each participant is enrolled in the study for 7 months, and 26 persons are randomized to one of the following 3 groups:

* Group 1; no intervention, observation with the OURA ring.
* Group 2: 12 weeks of physical activity guidance with short discussions via digital meetings regularly. They will conduct at least 150 minutes per week of moderate-intensity exercises. Brisk walks are the primary choice of activity; alternatively, swimming, cycling, or dancing to the physical exertion according to the Borg scale can be performed.
* Group 3: 12 weeks of sleep exercises. The lifestyle intervention of sleep will be delivered via an online group, with recommended home practices between sessions. Topics covered will include sleep education, sleep hygiene, and practices to improve sleep quality.

The study is digital and will use the platform "minforskning.se", which is validated according to GCP-GAMP5 and has the potential to collect digital consent forms.

ELIGIBILITY:
Inclusion Criteria:

* The MG disease status must be stable for at least six months before entry into the study; thus, the duration of the disease must be at least six months.
* Both patients with ocular and generalized MG are allowed to participate.
* For practical reasons, participants need to be able to understand fully and communicate in Swedish.

Exclusion Criteria:

* Participation in another clinical trial in the past 6 months.
* Disease duration less than 6 months.
* Contraindications to physical activity: unstable coronary syndrome or myocardial infarction within the preceding three months, respiratory failure (vital capacity < 70% predicted value) or cardiac failure (ejection fraction < 50% predicted value), concomitant neuromuscular diseases, disabling rheumatological disease (> 80% disability on the Barthel scale), chronic pain or disabling orthopedic conditions, hospitalization in the last three months for a serious medical or surgical condition, anemia (hematocrit < 30%), stroke within the previous year.
* MG patients already performing moderate-intensity physical activity of 150min or more per week, i.e., one of the target interventions.
* Pregnancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Myasthenia Gravis-Activities of Daily Living (MG-ADL) | 7 months
  Subjective assessment of MG-related fatiguability. A person's score can range from zero (normal) to 24 (most severe).

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | 7 months
  The Fatigue Severity Scale (FSS) ranges from 0 (least fatigue) to 63 (maximum fatigue).
Chalder Fatigue Scale | 7 months
  The Chalder Fatigue Scale ranges from 0 (least fatigue) to 33 (maximum fatigue)

OTHER OUTCOMES:
Heart rate variability | 7 months
  Heart rate variability is measured with the OURA ring.
Activity pattern | 7 months
  Number of steps and minutes in moderate and high intensity activity is measured by the OURA ring.
Percentage of deep sleep | 7 months
  The OURA ring measures the sleep stages, including time and percentage for deep sleep every night.
Circulating miRNA in serum | 7 months
  Changes in miR-150-5p and miR-30e-5p in serum samples.
Olink Target 96 Inflammation panel of cytokines | 7 months
  Changes in cytokine NPX protein values (log2 scaled) using Proximity Extension Assay (PEA) technology in serum samples

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rostedt Punga, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Not relevant.